CLINICAL TRIAL: NCT03138005
Title: Reduction of Oxygen After Cardiac Arrest (EXACT): The EXACT Study
Brief Title: Reduction of Oxygen After Cardiac Arrest
Acronym: EXACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic reduced enrolment and changed clinical protocols
Sponsor: Monash University (Other)
Collaborators: Ambulance Victoria (Other Government); SA Ambulance Service (Unknown); St John Ambulance Australia (Western Australia) (Unknown); Flinders University (Other); Curtin University (Other)
Responsible Party: Principal Investigator, Professor Stephen Bernard, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EXACT01; APP1107509 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2017-04-21; First posted 2017-05-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Emergency Care, Prehospital; Resuscitation; Oxygen; Cardiac Arrest; Heart Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- target SpO2 98-100% (Active Comparator): Post ROSC oxygen titrated to maintain SpO2 between 98-100%
  Interventions: Other: target SpO2 98-100%
- target SpO2 90-94% (Experimental): Post ROSC oxygen titrated to maintain SpO2 between 90-94%
  Interventions: Other: target SpO2 90-94%

INTERVENTIONS:
Other: target SpO2 98-100% — Prehospital, post-ROSC oxygen maintained at ≥10L/minute of oxygen (equivalent to ~100% oxygen) into SGA/ETT if hand ventilated or 100% (i.e. FiO2 of 1.0) oxygen settings if mechanically ventilated. Patients will continue on treatment to handover in the ED. Between arrival at ED and first ABG in ICU, the oxygen setting may then be decreased provided SpO2 is maintained between 98-100%.
  Arms: target SpO2 98-100%
Other: target SpO2 90-94% — Prehospital, post-ROSC oxygen reduced initially to 4L/minute (i.e. approximately 70% oxygen) into SGA/ETT if hand ventilated or an air mix setting if mechanically ventilated. If oxygen saturation remains ≥94% for 5 minutes, the oxygen flow rate will be further reduced to 2L/minute (i.e. approximately 46% oxygen) and hand ventilated to target an oxygen saturation between 90-94%. This treatment will continue to patient handover in the emergency department. Between arrival at ED and first ABG in ICU, oxygen will be titrated to target a oxygen saturation of 90-94%.
  Arms: target SpO2 90-94%

SUMMARY:
The Reduction of oxygen after cardiac arrest (EXACT) is a multi-centre, randomised, controlled trial (RCT) to determine whether reducing oxygen administration to target an oxygen saturation of 90-94%, compared to 98-100%, as soon as possible following successful resuscitation from OHCA improves outcome at hospital discharge.

DETAILED DESCRIPTION:
Currently out-of-hospital cardiac arrest (OHCA) patients who achieve ROSC are routinely ventilated with the highest fraction of inspired oxygen (FiO2) possible (i.e. FiO2 1.0 or 100% oxygen) until admission to an intensive care unit (ICU) - usually a period of 2 to 6 hours post-ROSC.

Post-ROSC oxygen therapy begins in the field by emergency medical services (EMS). EMS typically deliver a high flow of oxygen at rate of >10L/min (~100% oxygen), and use a pulse oximeter to monitor oxygen levels (SpO2). Normal SpO2 levels are considered to be 94% to 100%. The delivery of 100% oxygen is then usually continued throughout a patient's stay in the emergency department (ED) and during any diagnostic testing (e.g. computed tomography scans and cardiac angiography). During this time, oxygen is delivered to patients who remain unconscious via a mechanical ventilator, with levels continuously monitored by pulse oximetry and periodically by a blood test called an arterial blood gas (ABG). The ABG measurements include the oxygen pressure in the blood (PaO2) in mmHg. Once a patient is admitted to the ICU, the PaO2 is assessed and the oxygen fraction is typically reduced and then titrated (reduced or increased) on the ventilator to achieve a normal level of PaO2 ("normoxia") of between 80-100mmHg.

The administration of 100% oxygen for the first hours after resuscitation is based largely on convention and not on any supportive clinical data. It has been thought that maximizing oxygen delivery for several hours might be beneficial in a patient who has suffered profound deprivation of oxygen supply ("hypoxia") during a cardiac arrest. In addition, if a lower fraction of inspired oxygen is delivered, there is a perceived risk that the patient might become hypoxic (i.e. SpO2 <90% or PaO2 <80mmHg). Until recently, there has been no particular reason to recommend a decrease in oxygen delivery to the post-arrest patient prior to admission to ICU.

However, recent systematic reviews of compelling experimental data and supportive human observational studies indicate that the administration of 100% oxygen can create "hyperoxic" levels in the early post arrest period which may lead to additional neurological injury, and thus result in worse clinical outcome. No randomised control trials have yet tested titrating oxygen administration to lower but normal levels (i.e. "normoxia").

EXACT is a Phase 3 multi-centre, randomised, controlled trial (RCT) aiming to determine whether reducing oxygen administration to target an oxygen saturation of 90-94%, compared to 98-100%, as soon as possible following successful resuscitation from OHCA improves outcome at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years or older)
* Out-of-hospital cardiac arrest of presumed cardiac cause
* All cardiac arrest rhythms
* Unconscious (Glasgow Coma Scale <9)
* Return of spontaneous circulation
* Pulse oximeter measures oxygen saturation at ≥95% with oxygen flow set at >10L/min or FiO2 at 100%
* Patient has an endotracheal tube (ETT) or supraglottic airway (SGA) (e.g. laryngeal mask airway -LMA) and is spontaneously breathing or ventilated
* Transport is planned to a participating hospital

Exclusion Criteria:

* Female who is known or suspected to be pregnant
* Dependent on others for activities of daily living (i.e. facilitated care or nursing home residents)
* "Not for Resuscitation" order or Advanced Care Directives in place
* Pre-existing oxygen therapy (i.e. for COPD)
* Cardiac arrest due to drowning, trauma or hanging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Survival to hospital discharge | At hospital discharge, participants will be followed for the duration of hospital stay, an expected average of 2-4 weeks
  Survival to hospital discharge

SECONDARY OUTCOMES:
Neurological outcome | At hospital discharge, participants will be followed for the duration of hospital stay, an expected average of 2-4 weeks
  Cerebral Performance Category score
Incidence of hypoxia (SpO2<90%) | Before ICU admission, an expected average of 4-6 hours
  Incidence of hypoxia (SpO2<90%)
Recurrent cardiac arrest | Before ICU admission, an expected average of 4-6 hours
  Recurrent cardiac arrest requiring chest compressions before admission to ICU and not related to withdrawal of life sustaining-treatment
Myocardial Injury | First 24 hours of hospital admission
  Median peak troponin
Survival to intensive care unit discharge | Intensive care discharge, an expected average of 7 days
  Survival to intensive care unit discharge
Length of ICU stay | Intensive care discharge, an expected average of 7 days
  Length of ICU stay
Length of hospital stay | At hospital discharge, participants will be followed for the duration of hospital stay, an expected average of 2-4 weeks
  Length of hospital stay
Cause of death during hospital stay | At hospital discharge, participants will be followed for the duration of hospital stay, an expected average of 2-4 weeks
  e.g. cardiogenic shock, re-arrest with no ROSC, treatment withdrawn -hypoxic brain injury, brain death
Quality of Life SF-12 | 12 months
  The SF-12 Health Survey (SF-12) is a 12-item questionnaire used to assess health outcomes from the patient's perspective.
Quality of Life EQ-5D-3L | 12 months
  Quality of life assessment using the EQ-5D-3L descriptive system that comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Neurological Function | 12 months
  Modified Rankin Score
Degree of recovery (GOS-E) | 12 months
  Extended Glasgow Outcome Scale
Survival at 12 months | 12 months
  Survival at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bernard, Principal Investigator — Ambulance Victoria
Locations (21):
- Australia (21):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - SA Ambulance Service, Adelaide, South Australia
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Western Health: Footscray Hospital, Melbourne, Victoria
  - Western Health: Sunshine Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincents Hospital, Melbourne, Victoria
  - Northern Health: The Northern Hospital, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Ambulance Victoria, Melbourne, Victoria
  - Eastern Health: Maroondah Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Peninusla Health: Frankston Hospital, Melbourne, Victoria
  - Barwon Health: Geelong, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - St John Ambulance Western Australia, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] http://www.ambulance.vic.gov.au/Media/docs/VACAR-Annual-Report-201112-39a60ff4-083f-4893-af52-efeef570f6d1-0.pdf
- [Background] Kaneda T, Ku K, Inoue T, Onoe M, Oku H. Postischemic reperfusion injury can be attenuated by oxygen tension control. Jpn Circ J. 2001 Mar;65(3):213-8. doi: 10.1253/jcj.65.213. PMID 11266197
- [Background] Richards EM, Fiskum G, Rosenthal RE, Hopkins I, McKenna MC. Hyperoxic reperfusion after global ischemia decreases hippocampal energy metabolism. Stroke. 2007 May;38(5):1578-84. doi: 10.1161/STROKEAHA.106.473967. Epub 2007 Apr 5. PMID 17413048
- [Background] Pilcher J, Weatherall M, Shirtcliffe P, Bellomo R, Young P, Beasley R. The effect of hyperoxia following cardiac arrest - A systematic review and meta-analysis of animal trials. Resuscitation. 2012 Apr;83(4):417-22. doi: 10.1016/j.resuscitation.2011.12.021. Epub 2012 Jan 5. PMID 22226734
- [Background] Balan IS, Fiskum G, Hazelton J, Cotto-Cumba C, Rosenthal RE. Oximetry-guided reoxygenation improves neurological outcome after experimental cardiac arrest. Stroke. 2006 Dec;37(12):3008-13. doi: 10.1161/01.STR.0000248455.73785.b1. Epub 2006 Oct 26. PMID 17068310
- [Background] Saugstad OD. Resuscitation of newborn infants: from oxygen to room air. Lancet. 2010 Dec 11;376(9757):1970-1. doi: 10.1016/S0140-6736(10)60543-0. Epub 2010 Jul 19. No abstract available. PMID 20663546
- [Background] Hellstrom-Westas L, Forsblad K, Sjors G, Saugstad OD, Bjorklund LJ, Marsal K, Kallen K. Earlier Apgar score increase in severely depressed term infants cared for in Swedish level III units with 40% oxygen versus 100% oxygen resuscitation strategies: a population-based register study. Pediatrics. 2006 Dec;118(6):e1798-804. doi: 10.1542/peds.2006-0102. PMID 17142501
- [Background] Kilgannon JH, Jones AE, Shapiro NI, Angelos MG, Milcarek B, Hunter K, Parrillo JE, Trzeciak S; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Association between arterial hyperoxia following resuscitation from cardiac arrest and in-hospital mortality. JAMA. 2010 Jun 2;303(21):2165-71. doi: 10.1001/jama.2010.707. PMID 20516417
- [Background] Bellomo R, Bailey M, Eastwood GM, Nichol A, Pilcher D, Hart GK, Reade MC, Egi M, Cooper DJ; Study of Oxygen in Critical Care (SOCC) Group. Arterial hyperoxia and in-hospital mortality after resuscitation from cardiac arrest. Crit Care. 2011;15(2):R90. doi: 10.1186/cc10090. Epub 2011 Mar 8. PMID 21385416
- [Background] Ihle JF, Bernard S, Bailey MJ, Pilcher DV, Smith K, Scheinkestel CD. Hyperoxia in the intensive care unit and outcome after out-of-hospital ventricular fibrillation cardiac arrest. Crit Care Resusc. 2013 Sep;15(3):186-90. PMID 23944204
- [Background] Suzuki S, Eastwood GM, Glassford NJ, Peck L, Young H, Garcia-Alvarez M, Schneider AG, Bellomo R. Conservative oxygen therapy in mechanically ventilated patients: a pilot before-and-after trial. Crit Care Med. 2014 Jun;42(6):1414-22. doi: 10.1097/CCM.0000000000000219. PMID 24561566
- [Background] Kuisma M, Boyd J, Voipio V, Alaspaa A, Roine RO, Rosenberg P. Comparison of 30 and the 100% inspired oxygen concentrations during early post-resuscitation period: a randomised controlled pilot study. Resuscitation. 2006 May;69(2):199-206. doi: 10.1016/j.resuscitation.2005.08.010. Epub 2006 Feb 24. PMID 16500018
- [Background] Young P, Bailey M, Bellomo R, Bernard S, Dicker B, Freebairn R, Henderson S, Mackle D, McArthur C, McGuinness S, Smith T, Swain A, Weatherall M, Beasley R. HyperOxic Therapy OR NormOxic Therapy after out-of-hospital cardiac arrest (HOT OR NOT): a randomised controlled feasibility trial. Resuscitation. 2014 Dec;85(12):1686-91. doi: 10.1016/j.resuscitation.2014.09.011. Epub 2014 Sep 28. PMID 25261605
- [Background] Young P, Pilcher J, Patel M, Cameron L, Braithwaite I, Weatherall M, Beasley R. Delivery of titrated oxygen via a self-inflating resuscitation bag. Resuscitation. 2013 Mar;84(3):391-4. doi: 10.1016/j.resuscitation.2012.08.330. Epub 2012 Sep 3. PMID 22955052
- [Background] Bernard SA, Smith K, Cameron P, Masci K, Taylor DM, Cooper DJ, Kelly AM, Silvester W; Rapid Infusion of Cold Hartmanns Investigators. Induction of prehospital therapeutic hypothermia after resuscitation from nonventricular fibrillation cardiac arrest*. Crit Care Med. 2012 Mar;40(3):747-53. doi: 10.1097/CCM.0b013e3182377038. PMID 22020244
- [Background] Smith K, Andrew E, Lijovic M, Nehme Z, Bernard S. Quality of life and functional outcomes 12 months after out-of-hospital cardiac arrest. Circulation. 2015 Jan 13;131(2):174-81. doi: 10.1161/CIRCULATIONAHA.114.011200. Epub 2014 Oct 29. PMID 25355914
- [Background] Kenmure AC, Murdoch WR, Beattie AD, Marshall JC, Cameron AJ. Circulatory and metabolic effects of oxygen in myocardial infarction. Br Med J. 1968 Nov 9;4(5627):360-4. doi: 10.1136/bmj.4.5627.360. PMID 5683582
- [Background] Mak S, Azevedo ER, Liu PP, Newton GE. Effect of hyperoxia on left ventricular function and filling pressures in patients with and without congestive heart failure. Chest. 2001 Aug;120(2):467-73. doi: 10.1378/chest.120.2.467. PMID 11502645
- [Background] Nehme Z, Bernard S, Cameron P, Bray JE, Meredith IT, Lijovic M, Smith K. Using a cardiac arrest registry to measure the quality of emergency medical service care: decade of findings from the Victorian Ambulance Cardiac Arrest Registry. Circ Cardiovasc Qual Outcomes. 2015 Jan;8(1):56-66. doi: 10.1161/CIRCOUTCOMES.114.001185. PMID 25604556
- [Background] O'Driscoll BR, Howard LS, Davison AG; British Thoracic Society. BTS guideline for emergency oxygen use in adult patients. Thorax. 2008 Oct;63 Suppl 6:vi1-68. doi: 10.1136/thx.2008.102947. No abstract available. PMID 18838559
- [Background] Stub D, Bernard S, Duffy SJ, Kaye DM. Post cardiac arrest syndrome: a review of therapeutic strategies. Circulation. 2011 Apr 5;123(13):1428-35. doi: 10.1161/CIRCULATIONAHA.110.988725. No abstract available. PMID 21464058
- [Background] Neumar RW, Otto CW, Link MS, Kronick SL, Shuster M, Callaway CW, Kudenchuk PJ, Ornato JP, McNally B, Silvers SM, Passman RS, White RD, Hess EP, Tang W, Davis D, Sinz E, Morrison LJ. Part 8: adult advanced cardiovascular life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S729-67. doi: 10.1161/CIRCULATIONAHA.110.970988. PMID 20956224
- [Background] Soar J, Callaway CW, Aibiki M, Bottiger BW, Brooks SC, Deakin CD, Donnino MW, Drajer S, Kloeck W, Morley PT, Morrison LJ, Neumar RW, Nicholson TC, Nolan JP, Okada K, O'Neil BJ, Paiva EF, Parr MJ, Wang TL, Witt J; Advanced Life Support Chapter Collaborators. Part 4: Advanced life support: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2015 Oct;95:e71-120. doi: 10.1016/j.resuscitation.2015.07.042. Epub 2015 Oct 15. No abstract available. PMID 26477429
- [Derived] Bernard SA, Bray JE, Smith K, Stephenson M, Finn J, Grantham H, Hein C, Masters S, Stub D, Perkins GD, Dodge N, Martin C, Hopkins S, Cameron P; EXACT Investigators. Effect of Lower vs Higher Oxygen Saturation Targets on Survival to Hospital Discharge Among Patients Resuscitated After Out-of-Hospital Cardiac Arrest: The EXACT Randomized Clinical Trial. JAMA. 2022 Nov 8;328(18):1818-1826. doi: 10.1001/jama.2022.17701. PMID 36286192
- [Derived] Bray JE, Smith K, Hein C, Finn J, Stephenson M, Cameron P, Stub D, Perkins GD, Grantham H, Bailey P, Brink D, Dodge N, Bernard S; EXACT investigators. The EXACT protocol: A multi-centre, single-blind, randomised, parallel-group, controlled trial to determine whether early oxygen titration improves survival to hospital discharge in adult OHCA patients. Resuscitation. 2019 Jun;139:208-213. doi: 10.1016/j.resuscitation.2019.04.023. Epub 2019 Apr 19. PMID 31009695